CLINICAL TRIAL: NCT06312111
Title: Assessment of Physical Activity and Various Aspects of Quality of Life in Patients With Pulmonary Arterial Hypertension
Brief Title: Physical Activity and Various Aspects of Quality of Life in Patients With Pulmonary Arterial Hypertension (Ph-PAH)
Acronym: PhA-PAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62/2021
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Arterial Hypertension; Physical Inactivity
Keywords: pulmonary arterial hypertension; education; self-monitoring; physical activity; step count
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A physically inactive subgroup (Experimental): Patients who walked <5,000 steps per day during the first two weeks
  Interventions: Behavioral: recommendation to increase physical activity
- A physically active subgroup (Active Comparator): Patients who walked >5,000 steps per day during the first two weeks
  Interventions: Behavioral: recommendation to increase physical activity

INTERVENTIONS:
Behavioral: recommendation to increase physical activity — education on the benefits of physical activity in PAH from the first visit and doctor's recommendation to increase physical activity above 5,000 steps a day in inactive patients and above 5,000 steps per person in active patients

SUMMARY:
Evaluate whether education, a simple doctor's recommendation to increase physical activity in inactive patients, and self-monitoring of physical activity using a pedometer were effective and beneficial for patients with pulmonary arterial hypertension (PAH)

DETAILED DESCRIPTION:
Each patient was educated about the benefits of PhA in PAH on the initial visit. Patients wore pedometers (Omron HJ-321-E) for 2 weeks. After PhA assessment, the patients were contacted by a physician. Patients who walked <5,000 steps per day were recommended to increase PhA, and patients who walked ≥5,000 steps per day were recommended to maintain PhA. Patients wore pedometers for 3 months until their next visit. The primary endpoint was the number of steps after 12 weeks of the study; the secondary endpoint was the 6-minute walk test distance (6MWD), quality of life (SF-36), acceptance of the disease, and anxiety and depression level (HADS).

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years
* PAH diagnosis according to current guidelines, confirmed by right heart catheterization
* optimal pharmacological treatment
* stable clinical condition at least 3 months before inclusion in the study
* Informed consent to participate in your own

Exclusion Criteria:

* Age under 18 years
* a type of hypertension other than PAH
* a neurological or orthopedic disease that prevents walking and performing the 6-minute walk test
* mental illness that prevents cooperation and assessment of quality of life survey
* lack of consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2022-07-17 (Actual)

PRIMARY OUTCOMES:
Number of steps per day | At baseline, after initial period 2 weeks
  Number of steps per day monitored by pedometer Omron HJ-321-E

SECONDARY OUTCOMES:
Change in 6-minute walk distance | At baseline, 3 months
  Distance in six-minute walk test
Change in quality of life (SF-36) | At baseline, 3 months
  Change in quality of life recorded by patient questionnaire 36-Item Short Form Health Survey (SF-36)
Change in the hospital anxiety and depression scale (HADS) | At baseline, 3 months
  level of anxiety and depression measured by hospital anxiety and depression scale (HADS)
Change in the acceptance of illness (AIS) | At baseline, 3 months
  acceptance of illness measured by acceptance of illness scale (AIS)
Change in N-Terminal Pro-B-Type Natriuretic Peptide level (NT-proBNP) | At baseline, 3 months
  Blood sample to measure the concentration of N-terminal Pro-B type natriuretic peptide
Change in World Health Organization (WHO) functional Class recorded by investigator in conjunction with the 6MWD | At baseline, 3 months
  WHO functional class assessment
Compliance with counting steps | at 3 months
  Compliance with counting steps

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary Circulation, Thromboembolic Diseases and Cardiology, European Health Centre, Otwock, Centre of Postgraduate Medical Education, Otwock, Borowa 14/18, Poland

IPD SHARING:
Plan to Share IPD: No